CLINICAL TRIAL: NCT03943654
Title: Novel Approach to Improve Patient Care and Diarrheal Disease Research Using Mobile Technology
Brief Title: Improving Nighttime Access to Care and Treatment (Part 2)
Acronym: INACT2
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Universite d'Etat d'Haiti (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201802920 -N; DP5OD019893 (NIH)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Acute Diarrhea; Acute Respiratory Infection; Acute Febrile Illness
Keywords: Telemedicine; Diarrhea; Diarrhoea; mHealth; Healthline
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool samples and nasal swabs will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children living within study delivery area w/o danger signs: Families who call the healthline service about a sick child (no danger signs) and live within the mobile pharmacy delivery area will receive illness assessments and treatment recommendations over the phone. Immediately following calls a nurse will conduct household visits to complete in-person assessments of the children. Illness progression will be tracked with a 8-12 day follow up call. The phone and in-person assessments will be compared to evaluate safety and accuracy of the healthline.
  Interventions: Other: MotoMeds Healthline- illness assessment and treatment recommendation for non-emergent cases by telephone
- Children living outside study delivery area w/o danger signs: Families who call the healthline service about a sick child (no danger signs) and live outside the delivery area will receive illness assessments and treatment recommendations over the phone. Illness progression will be tracked with a 8-12 day follow up call.
  Interventions: Other: MotoMeds Healthline- illness assessment and treatment recommendation for non-emergent cases by telephone
- Children who are identified as having danger signs: Families who call the healthline service about a sick child and who are identified as having a danger sign will be directed to the nearest medical facility. Illness progression will be tracked with a 8-12 day follow up call.
  Interventions: Other: MotoMeds Healthline- illness assessment and treatment recommendation for non-emergent cases by telephone

INTERVENTIONS:
Other: MotoMeds Healthline- illness assessment and treatment recommendation for non-emergent cases by telephone — The healthline uses a series of questions (based off of the WHO Integrated Management of Childhood Illness guidelines) asked to the parent of a sick child over the phone to remotely triage and assess the child's illness and then provide a treatment recommendation. MotoMeds is the accompanying motorcycle delivery service for basic medication delivery at nighttime.

SUMMARY:
Children in resource-limited settings who develop illness at night are often isolated from pre-emergency care, resulting in progression to an emergency because families are forced to wait until morning to seek care. This is especially true in Haiti based on needs assessments (INACT Part 1; INACT1) surrounding access to healthcare. This study (INACT Part 2; INACT2) seeks to improve access to care by establishing a health hotline (healthline) and mobile pharmacy for families with children who become ill at nighttime. The healthline will be staffed by medical professionals and will provide phone based assessment and treatment recommendations based on standard of care practices according to Haitian and WHO guidelines. The healthline will focus on pre-emergency patients (those without danger signs as defined by WHO guidelines). Emergent patients will be advised to bypass the healthline and seek immediate care at the nearest medical facility. In the event that a non-emergent patient requires access to basic medications or fluids and is logistically accessible, the mobile pharmacy service will be offered.

The specific aims of the study are as follows: Aim I. Evaluate congruence between healthline assessment over the phone and in-person assessment of participants (patients using the healthline) 10 years of age and younger. The investigators hypothesize that in-person assessments based on WHO guidelines will be discordant with those made by the healthline because the physical aspects of the call-center assessment will be performed by an untrained parent/ guardian. The study focuses on acute diarrheal disease (ADD) and acute respiratory illness (ARI) but is not exclusive to these two chief complaints. Aim II: Identify determinants that correlate with seeking care at a medical facility over the 8-12 day follow up period after the initial call. The findings from this study will determine if a healthline model is a safe and accurate method of providing high quality access to nighttime healthcare, averting the progression of non-emergent cases to emergencies.

ELIGIBILITY:
Inclusion Criteria:

* age of patient must be 10 years or younger
* patient must reside inside the study delivery area
* consent/assent to participate

Exclusion Criteria:

* emergent illness (danger signs present)

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The healthine service will be advertised to residents in or approximate to a 5Km radius centered around the healthline office, which is in the community of La Reserve, Gressier, Haiti. There are approximately 12,632 households in this area covering 79 sq km.
Sampling Method: Non-Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Congruence between phone and in person clinical assessment. | Begins when the healthline call is placed and ends once the nurse has completed the household visit; approximately 1-3 hours.
  The responses parents give over the phone describing the child's illnesses will be compared to the routine clinical exam that the nurse performs in person. Clinical assessment features include vital signs, signs of work of breathings, and signs of dehydration per WHO and APP guidelines.

SECONDARY OUTCOMES:
Determinants that correlate with seeking care at a medical facility | Begins when the healthline call is placed and ends 8-12 days later.
  A follow up call will be placed 8-12 days after the initial healthline call to investigate factors associated with seeking care at a medical facility after the initial call to the heathline service.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Nelson, MD PHD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Public Health Research Laboratory, Gressier, Ouest, Haiti

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klarman MB, Chi X, Cajusma Y, Flaherty KE, Capois AC, Dofine MDV, Exantus L, Friesen J, Beau de Rochars VM, Becker T, Baril C, Gurka MJ, Nelson EJ. Development and evaluation of a clinical guideline for a paediatric telemedicine service in a low-resource setting. BMJ Paediatr Open. 2024 Jan 8;8(1):e002164. doi: 10.1136/bmjpo-2023-002164. PMID 38191203
- [Derived] Klarman MB, Flaherty KE, Chi X, Cajusma Y, Capois AC, Vladimir Dofine MD, Exantus L, Friesen J, Beau de Rochars VM, Baril C, Gurka MJ, Becker TK, Nelson EJ. Implementation of a Pediatric Telemedicine and Medication Delivery Service in a Resource-limited Setting: A Pilot Study for Clinical Safety and Feasibility. J Pediatr. 2023 Jun;257:113304. doi: 10.1016/j.jpeds.2022.12.005. Epub 2022 Dec 14. PMID 36528053
- See also: Eric Nelson Research Program at UF — https://nelson.research.pediatrics.med.ufl.edu